CLINICAL TRIAL: NCT02265848
Title: Single Blinded, Randomized Control Trial of High Frequency Stimulation in Subjects With Precision® Spinal Cord Stimulator System to Assess Efficacy and Preferability in Back and Extremity Pain Relief
Brief Title: High Frequency Stimulation Trials in Patients With Precision Spinal Cord Stimulator System
Acronym: HFSCS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Center for Clinical Research, Winston-Salem, NC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IIR-2014-01
Record Dates: First submitted 2014-09-30; First posted 2014-10-16 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Pain; Low Back Pain; Radiculopathy; Complex Regional Pain Syndrome (CRPS)
Keywords: Spinal cord stimulation; Chronic pain; Chronic low back pain; Radiculopathy; Complex Regional Pain Syndrome (CRPS); High Frequency stimulation
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Radiculopathy; Complex Regional Pain Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group A (Active Comparator): Subjects assigned to treatment group A will begin the 7 week study with high frequency stimulation for first 3 weeks of the study. After first 3 weeks, subject will return to clinic to turn off the SCS device, and will start 7-10 days of wash off period. At the end of the wash off period, subject will return to clinic and have the SCS device turned on to have it programmed to deliver the low frequency stimulation for the next 3 weeks. At the end of the 7th week, the subject will return for final end of treatment visit for conclusion of the study.
  Interventions: Other: High frequency stimulation; Other: Low frequency stimulation
- Treatment group B (Active Comparator): Subjects assigned to treatment group B will begin the 7 week study with low frequency stimulation for first 3 weeks of the study. After first 3 weeks, subject will return to clinic to turn off the SCS device, and will start 7-10 days of wash off period. At the end of the wash off period, subject will return to clinic and have the SCS device turned on to have it programmed to deliver the high frequency stimulation for the next 3 weeks. At the end of the 7th week, the subject will return for final end of treatment visit for conclusion of the study.
  Interventions: Other: High frequency stimulation; Other: Low frequency stimulation

INTERVENTIONS:
Other: High frequency stimulation — Implanted pulse generator of a spinal cord stimulator will programmed to deliver high frequency stimulation for pain relief. For our purposes, high frequency stimulation will be defined as 1000 hertz.
Other: Low frequency stimulation — Implanted pulse generator of a spinal cord stimulator will programmed to deliver low frequency stimulation for pain relief. Low frequency stimulation will be defined as conventional stimulation pulse generator programming.

SUMMARY:
Study designed to compare the conventional stimulation programming versus the high frequency stimulation programming of the spinal cord stimulator for subjects who already have a spinal cord stimulator.

DETAILED DESCRIPTION:
Subject with Precision models of spinal cord stimulators will be invited to take part in the study that will compare the high frequency stimulation versus low frequency stimulation to look for any changes in efficacy, and preferability between high and low frequency stimulation program for the spinal cord stimulator (SCS) system.

The study is designed as 7 week study that can take up to 9 weeks per subject. 7 weeks are divided into 3 segments. First segment will be 3 weeks of spinal cord stimulation followed by second segment of wash off period, which will take 1 week (7 days), then the last segment with 3 weeks of spinal cord stimulation. At the end of each segments, there will be a follow up visits.

Each follow up visits can occur up to 5 business days after the follow up due date for post spinal cord stimulation follow ups, and up to 3 business days after the follow up due date for the post wash off visit.

At each visits, including baseline, subject will be asked to answer Numeric Pain Rating Scale (NPRS), Oswestry Disability Index (ODI), and Patients Global Impression of Change (PGIC) to assess interval effect of the programming parameter for the spinal cord stimulator.

Visit schedule and assessment summary:

Visit 1: Screening and Baseline

* Review inclusion and exclusionary criteria (I&E)
* Informed Consent
* Demographics, Medical History
* Physical examination, Vital signs.
* Randomization (A, or B) and programming of devices according to randomization
* Baseline questionnaires
* Numeric Pain Rating Scale (NPRS) to measure the pain experienced by the subject over 1 week prior to enrolling in the study. this will include best pain, worse pain, and average pain as well as pain at the time of enrollment.
* Oswestry disability index (ODI) will measure the average disability caused by the painful condition approximately 3 weeks prior to the enrollment in to the study. Subject will be asked on 10 different categories of activities of daily living. They are: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling.
* Patients Global Impression of Change (PGI-C) will be asked to assess the subject's impression of their painful condition, since the implanting of the spinal cord stimulator.
* Concomitant medications

Visit 2: (end of 3 week assessments, + 5 days) End of first treatment period

* Interim Questionnaires:
* NPRS: We will measure pain experienced by the subject over 3 weeks since the last research visit (visit 1),prior to visit 2. This will include best pain, worse pain, and average pain as well as pain at the time of enrollment.
* Oswestry disability index will measure the disability caused by the painful condition since last visit of the study (visit 1), which covers 3 weeks of duration after the last research visit. Subject will be asked on 10 different categories of activities of daily living. They are: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling.
* PGI-C will be asked to assess the subject's impression of their painful condition, since the last visit of the study (visit 1), which covers 3 weeks of duration since the last research visit, prior to visit 2.
* Device Interrogation and turn off SCS for 7 to 10 days
* Start wash off period for 7 to 10 days
* Review Adverse Events (AE) and Concomitant medications (Con meds)

Visit 3: (end of wash off period, +3 days) Beginning of second treatment period

* Questionnaires:
* NPRS to measure the pain experienced by the subject over 1 week since visit 2, prior to visit 3, this will include best pain, worse pain, and average pain as well as pain at the time of enrollment.
* Oswestry disability index will measure the disability caused by the painful condition 1 week since last visit 2, prior to the visit 3. Subject will be asked on 10 different categories of activities of daily living. They are: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling.
* PGI-C will be asked to assess the subject's impression of their painful condition, during the last 1 week since visit 2, prior to visit 3.
* Device interrogation and programming; start of next treatment period.
* Review AE and Con meds.

Visit 4: (end of 3 week assessment +5 days) End of Treatment

* End of second treatment period.
* End of treatment Questionnaires:
* NPRS: We will measure pain experienced by the subject over 3 weeks since the last research visit (visit 3) prior to visit 4. This will include best pain, worse pain, and average pain as well as pain at the time of enrollment.
* Oswestry disability index will measure the disability caused by the painful condition since last visit of the study, which covers 3 weeks of duration after the last research visit (visit 3). Subject will be asked on 10 different categories of activities of daily living. They are: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling.
* PGI-C will be asked to assess the subject's impression of their painful condition, since the last visit of the study, which covers 3 weeks of duration since the last research visit (visit 3), prior to visit 4.
* Device Interrogation and re-programming if necessary.
* Review AE's and Con meds

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years and older, and younger than 70 years of age.
2. Subject has had a Precision® spinal cord stimulator system implanted for chronic painful condition.
3. Subject pain scores >5 on NPRS

Exclusion Criteria:

1. Currently diagnosed with cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to assess pain
2. Unstable medical or psychiatric illness
3. Lifetime history of psychosis, hypomania, or mania.
4. Epilepsy, or dementia
5. Substance abuse in the last 6 months
6. Pregnant or breastfeeding
7. Not on contraception for those of childbearing age. (Barrier methods, oral contraception, hormone injections, or surgical sterilization)
8. Treatment with investigational drug within 30 days of screening.
9. Concomitant medication exclusions consisting of medications or herbal agents with central nervous system (CNS) effects with exception of episodic use of sedating antihistamines

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M North, MD, Principal Investigator — The Carolinas Pain Institute
Locations (1):
- Center for Clinical Research, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No individual participants data will be shared with anyone other than study staff for analysis purposes.

REFERENCES:
- [Background] Simpson BA. Spinal cord stimulation. Br J Neurosurg. 1997 Feb;11(1):5-11. doi: 10.1080/02688699746627. No abstract available. PMID 9156011
- [Background] Lee D, Hershey B, Bradley K, Yearwood T. Predicted effects of pulse width programming in spinal cord stimulation: a mathematical modeling study. Med Biol Eng Comput. 2011 Jul;49(7):765-74. doi: 10.1007/s11517-011-0780-9. Epub 2011 Apr 29. PMID 21528381
- [Background] Kemler MA, Barendse GA, van Kleef M, de Vet HC, Rijks CP, Furnee CA, van den Wildenberg FA. Spinal cord stimulation in patients with chronic reflex sympathetic dystrophy. N Engl J Med. 2000 Aug 31;343(9):618-24. doi: 10.1056/NEJM200008313430904. PMID 10965008
- [Background] Gordon AT, Zou SP, Kim Y, Gharibo C. Challenges to setting spinal cord stimulator parameters during intraoperative testing: factors affecting coverage of low back and leg pain. Neuromodulation. 2007 Apr;10(2):133-41. doi: 10.1111/j.1525-1403.2007.00101.x. PMID 22151862
- [Background] Wu M, Linderoth B, Foreman RD. Putative mechanisms behind effects of spinal cord stimulation on vascular diseases: a review of experimental studies. Auton Neurosci. 2008 Feb 29;138(1-2):9-23. doi: 10.1016/j.autneu.2007.11.001. PMID 18083639
- [Background] Fisher LE, Tyler DJ, Triolo RJ. Optimization of selective stimulation parameters for multi-contact electrodes. J Neuroeng Rehabil. 2013 Feb 27;10:25. doi: 10.1186/1743-0003-10-25. PMID 23442372
- [Background] Guan Y, Wacnik PW, Yang F, Carteret AF, Chung CY, Meyer RA, Raja SN. Spinal cord stimulation-induced analgesia: electrical stimulation of dorsal column and dorsal roots attenuates dorsal horn neuronal excitability in neuropathic rats. Anesthesiology. 2010 Dec;113(6):1392-405. doi: 10.1097/ALN.0b013e3181fcd95c. PMID 21068658
- [Background] El-Khoury C, Hawwa N, Baliki M, Atweh SF, Jabbur SJ, Saade NE. Attenuation of neuropathic pain by segmental and supraspinal activation of the dorsal column system in awake rats. Neuroscience. 2002;112(3):541-53. doi: 10.1016/s0306-4522(02)00111-2. PMID 12074897
- [Background] Cui JG, O'Connor WT, Ungerstedt U, Linderoth B, Meyerson BA. Spinal cord stimulation attenuates augmented dorsal horn release of excitatory amino acids in mononeuropathy via a GABAergic mechanism. Pain. 1997 Oct;73(1):87-95. doi: 10.1016/s0304-3959(97)00077-8. PMID 9414060
- [Background] Cui JG, Meyerson BA, Sollevi A, Linderoth B. Effect of spinal cord stimulation on tactile hypersensitivity in mononeuropathic rats is potentiated by simultaneous GABA(B) and adenosine receptor activation. Neurosci Lett. 1998 May 15;247(2-3):183-6. doi: 10.1016/s0304-3940(98)00324-3. PMID 9655623
- [Background] Song Z, Meyerson BA, Linderoth B. The interaction between antidepressant drugs and the pain-relieving effect of spinal cord stimulation in a rat model of neuropathy. Anesth Analg. 2011 Nov;113(5):1260-5. doi: 10.1213/ANE.0b013e3182288851. Epub 2011 Jul 25. PMID 21788322
- [Background] Song Z, Meyerson BA, Linderoth B. Spinal 5-HT receptors that contribute to the pain-relieving effects of spinal cord stimulation in a rat model of neuropathy. Pain. 2011 Jul;152(7):1666-1673. doi: 10.1016/j.pain.2011.03.012. Epub 2011 Apr 22. PMID 21514998
- [Background] Ding X, Hua F, Sutherly K, Ardell JL, Williams CA. C2 spinal cord stimulation induces dynorphin release from rat T4 spinal cord: potential modulation of myocardial ischemia-sensitive neurons. Am J Physiol Regul Integr Comp Physiol. 2008 Nov;295(5):R1519-28. doi: 10.1152/ajpregu.00899.2007. Epub 2008 Aug 27. PMID 18753268
- [Background] Smits H, van Kleef M, Joosten EA. Spinal cord stimulation of dorsal columns in a rat model of neuropathic pain: evidence for a segmental spinal mechanism of pain relief. Pain. 2012 Jan;153(1):177-183. doi: 10.1016/j.pain.2011.10.015. Epub 2011 Nov 9. PMID 22078661
- [Background] Prager JP. What does the mechanism of spinal cord stimulation tell us about complex regional pain syndrome? Pain Med. 2010 Aug;11(8):1278-83. doi: 10.1111/j.1526-4637.2010.00915.x. PMID 20704677
- [Background] Buonocore M, Bodini A, Demartini L, Bonezzi C. Inhibition of somatosensory evoked potentials during spinal cord stimulation and its possible role in the comprehension of antalgic mechanisms of neurostimulation for neuropathic pain. Minerva Anestesiol. 2012 Mar;78(3):297-302. PMID 22095108
- [Background] Parker JL, Karantonis DM, Single PS, Obradovic M, Cousins MJ. Compound action potentials recorded in the human spinal cord during neurostimulation for pain relief. Pain. 2012 Mar;153(3):593-601. doi: 10.1016/j.pain.2011.11.023. Epub 2011 Dec 19. PMID 22188868
- [Background] Ito S, Sugiura T, Azami T, Sasano H, Sobue K. Spinal cord stimulation for a woman with complex regional pain syndrome who wished to get pregnant. J Anesth. 2013 Feb;27(1):124-7. doi: 10.1007/s00540-012-1462-y. Epub 2012 Aug 15. PMID 23011119
- [Background] Yoo HS, Nahm FS, Yim KH, Moon JY, Kim YS, Lee PB. Pregnancy in woman with spinal cord stimulator for complex regional pain syndrome: a case report and review of the literature. Korean J Pain. 2010 Dec;23(4):266-9. doi: 10.3344/kjp.2010.23.4.266. Epub 2010 Dec 1. PMID 21217892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All study subjects were recruited from the Carolinas Pain Institute who were implanted with Boston Scientific's Precision Plus spinal cord stimulation (SCS) system for chronic axial pain, and at the time of recruitment, was not receiving adequate pain relief from SCS system with baseline numeric pain rating scale of 5 or greater.
Pre-assignment Details: Randomization scheme was 1 to 1 ratio. Randomization assignment was generated using random number generator, and individual results were sealed in an envelope. If subject needed to be replaced, the replacement subject will receive the same randomization assignment.
Groups:
- Treatment Group A: Subjects randomized to the treatment group A will begin the 7 week study "per sequence" (e.g., "High frequency first, then Low frequency" and "Low frequency first, then High frequency"), with each stimulation modes lasting approximately 3 weeks with 7 to 10 days of "wash off" periods in between. At the end of the 7th week, the subject will return for final end of treatment visit for conclusion of the study.
- Treatment Group B: Subjects randomized to the treatment group B will begin the 7 week study "per sequence" (e.g., "Low frequency first, then High frequency" and "High frequency first, then Low frequency"), with each stimulation modes lasting approximately 3 weeks with 7 to 10 days of "wash off" periods in between. At the end of the 7th week, the subject will return for final end of treatment visit for conclusion of the study.
Period: Overall Study
Arm/Group | Treatment Group A | Treatment Group B
Started | 11 (First subject for this study was randomized on October 1st 2014) | 11
Completed | 11 | 11 (Last subject for this study completed the visit on December 24, 2014)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group A: Subjects randomized to the treatment group A will begin the 7 week study with high frequency (1000Hz) sub-perception stimulation for first 3 weeks of the study. After first 3 weeks, subject will return to clinic to turn off the SCS device, and will start 7-10 days of wash off period. At the end of the wash off period, subject will return to clinic and have the SCS device turned on to have it programmed to deliver the low frequency stimulation for the next 3 weeks. At the end of the 7th week, the subject will return for final end of treatment visit for conclusion of the study.
- Treatment Group B: Subjects randomized to the treatment group B will begin the 7 week study with low frequency (40 to 50Hz) paresthesia capture stimulation for first 3 weeks of the study. After first 3 weeks, subject will return to clinic to turn off the SCS device, and will start 7-10 days of wash off period. At the end of the wash off period, subject will return to clinic and have the SCS device turned on to have it programmed to deliver the high frequency (1000Hz) sub-perception stimulation for the next 3 weeks. At the end of the 7th week, the subject will return for final end of treatment visit for conclusion of the study.
- Total: Total of all reporting groups
Arm/Group | Treatment Group A | Treatment Group B | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 59 [45 to 75] | 56 [36 to 72] | 57 [36 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: Digital pain rating system that scores patient's subjective pain rating from 0 to 10; with greater number indicating progressively worsening pain. NPRS were measured at baseline (visit1), and at each follow ups visits at visit 2, 3 and 4. Visit 2 and 4 captured post treatment (either 1000 Hz or standard stimulation depending on the randomization) results, and visit 3 captured NPRS after the wash off from the spinal cord stimulation.
Time Frame: Baseline (visit 1), and at each follow up visits (visits 2, 3, and 4)
Population: All study subjects were implanted with Boston Scientific's Precision Plus spinal cord stimulation system for treatment of chronic axial pain.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 11 | 11
units on a scale
  Average Baseline NPRS Score | 6.09 [3 to 10] | 6.27 [4 to 8]
  Average NPRS after 1000 Hz. stimulation | 3.73 [1 to 8] | 3.82 [1 to 6]
  Average NPRS after standard stimulation | 5.64 [4 to 8] | 6.09 [4 to 8]
  Average NPRS after Wash off | 6.45 [4 to 10] | 7.18 [4 to 9]
  Best Baseline NPRS score | 3.72 [1 to 7] | 4.45 [2 to 7]
  Best NPRS score after 1000 Hz. stimulation | 2.64 [1 to 8] | 2.18 [1 to 6]
  Best NPRS score after standard stimulation | 3.46 [1 to 6] | 4.45 [2 to 7]
  Best NPRS after Wash off | 4.54 [2 to 9] | 5.36 [1 to 8]
  Worst Baseline NPRS score | 7.90 [6 to 10] | 8.09 [5 to 10]
  Worst NPRS score after 1000 Hz. stimulation | 6.64 [3 to 9] | 6.64 [3 to 10]
  Worst NPRS score after standard stimulation | 8.18 [5 to 10] | 8.36 [6 to 10]
  Worst NPRS after Wash off | 8.72 [6 to 10] | 8.81 [7 to 10]

2. Secondary Outcome: Oswestry Disability Index Questionnaire (ODI).
Description: ODI is a outcome metrics that is design to assess the severity of disability based on 10 activity categories. ODI is based on 0 to 100% scale, where larger percentage implies worse disability. (There are 5 categories: 0-20%: Minimal disability, 21-40%: Moderate disability, 41-60%: Severe disability, 61-80%: Crippled. 81-100%: Either bed bound or exaggerating symptoms). ODI were measured at baseline (visit1), and at each follow ups visits at visit 2, 3 and 4. Visit 2 and 4 captured post treatment (either 1000 Hz or standard stimulation depending on the randomization) results, and visit 3 captured NPRS after the wash off from the spinal cord stimulation.
Time Frame: Baseline (visit 1), and at each follow up visits (visits 2, 3, and 4)
Population: as for outcome 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 11 | 11
units on a scale
  Baseline ODI score | 47.49 [24 to 68] | 51.25 [36 to 60]
  ODI after 1000 Hz. stimluation | 39.23 [24 to 66] | 33.77 [16 to 54]
  ODI after standard stimulation | 49.63 [28 to 70] | 49.05 [30 to 58]
  ODI after wash off | 52.87 [20 to 76] | 56.77 [32 to 78]

3. Secondary Outcome: Patient's Global Impression of Change (PGIC)
Description: PGIC is a 7-point scale that requires study subjects to rate the severity of their illness or medical condition after a specific treatment. 1: No change, 2: Almost the same, 3: A little better, 4: Somewhat better, 5: Moderately better, 6: Better, 7: A great deal better. Study subjects were asked to report their impression of changes at baseline visit, visit 2 through 4.
Time Frame: Baseline (visit 1), and at each follow up visits (visits 2, 3, and 4)
Population: as for outcome 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 11 | 11
units on a scale
  PGIC After 1000 Hz. stimulation | 4.27 [3 to 6] | 5.91 [4 to 7]
  PGIC after standard stimulation | 2.54 [1 to 7] | 2.45 [1 to 6]
  PGIC after Wash off | 1.45 [1 to 3] | 1.27 [1 to 2]

4. Other Pre Specified Outcome: Preferability
Description: At the conclusion of the study, subjects were asked to report which spinal cord stimulation modes they preferred. Subjects were presented with two boxes (1000 Hz. stimulation and Standard stimulation) and asked to check one.
Time Frame: End of treatment visit on visit 4
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 11 | 11
participants
  Subjects who prefer 1000 Hz. stimulation | 8 | 10
  Subjects who prefer standard stimulation | 3 | 1

ADVERSE EVENTS:
Time Frame: All adverse events, including serious adverse events were collected during the study duration. First study subject was enrolled on October 1st of 2014, and last subjects completed the scheduled visit on December 24 of 2014.
Description: If adverse events or serious adverse events were reported during the study duration, study staff and principal investigator were to follow the adverse event until the resolution. However, there were no adverse events reported during the study duration, thus no subjects were followed beyond study duration.
Arm/Group | Treatment Group A | Treatment Group B
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
This study was limited by the sampling size, and by device type. Study was open to subjects who were implanted with Boston Scientific's Precision Plus device only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No